CLINICAL TRIAL: NCT05413083
Title: Dynamic Assessment of Cardiac Function in Acutely Decompensated Cirrhosis
Brief Title: Evaluation of Cardiac Function in Acutely Decompensated Cirrhosis
Acronym: DYNACORD-AD
Status: Active, not recruiting | Type: Observational
Sponsor: Clinical Hospital Colentina (Other)
Responsible Party: Principal Investigator, Andrei Voiosu, Principal investigator, Clinical Hospital Colentina
Other Study IDs: DYNACORD-AD
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Cirrhosis; Acute Liver Failure; Cardiomyopathies
MeSH Terms: conditions — Fibrosis; Liver Failure, Acute; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples Without DNA — centrifuged serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to investigate cardiac function in patients with cirrhosis in the acute setting. Acute decompensation and acute-on-chronic liver failure are major events in the life of a patient as they herald disease progression and negative prognosis. Cardiocirculatory function will be assessed by serial assessments in patients admitted for acute decompensation of cirrhosis.

DETAILED DESCRIPTION:
In this project we aim to investigate the dynamic role of cardiac function in the short-term evolution of patients with AD of cirrhosis through noninvasive and accessible tests and validate prognostic imaging and serum biomarkers. The main objectives are:

1. To describe changes and evolution of cardiac function in AD of cirrhosis
2. To investigate associations between echocardiographic parameters and serum biomarkers
3. To investigate the association between ACLF and cardiac dysfunction
4. To assess the short-term prognostic impact of cardiac function in AD and ACLF;
5. To evaluate the added predictive value of cardiac markers to current scores (CLIF-C).

ELIGIBILITY:
Inclusion Criteria:

* proven cirrhosis with acute decompensation

Exclusion Criteria:

* screening after > 72 hours from admission
* previous severe cardiac conditions (e.g. ischemic heart disease, atrial fibrillation, congestive heart failure, ICD)
* concomitant severe disease (e.g. active neoplasia, severe COPD, etc)
* lack of informed consent
* intubated/ comatose patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cirrhotic patients admitted for acute decompensated cirrhosis will be screened, regardless of gender, etiology of liver disease, and age (if above 18 years).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
cardiac dysfunction | 90 days
  rate of onset and evolution of systolic/ diastolic dysfunction in acute decompensation
composite outcome | 90 days
  risk of developing ACLF, disease worsening, or death during follow-up

SECONDARY OUTCOMES:
biomarkers | 30 days
  detecting biomarkers predictive for cardiac dysfunction and disease severity

CONTACTS AND LOCATIONS:
Locations (1):
- Spitalul clinic Colentina, Bucharest, Romania